CLINICAL TRIAL: NCT02256046
Title: Predictive Factors and Outcome of Esophageal Ulcers After Endoscopic Treatment of Esophageal Varices; Multicenter Study
Brief Title: Predictive Factors and Outcome of Esophageal Ulcers After Endoscopic Treatment of Esophageal Varices
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ibrahim Shebl, Dr., Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: esophageal ulcers
Record Dates: First submitted 2014-09-26; First posted 2014-10-03 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Esophageal and Gastric Varices; Ulcer; Cirrhosis; Hypertension, Portal
MeSH Terms: conditions — Esophageal and Gastric Varices; Ulcer; Fibrosis; Hypertension, Portal | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Esophagogastroduodenoscope (Experimental): Endoscopic therapies for varices aim to reduce variceal wall tension by obliteration of the varix. The two principal methods available for esophageal varices are endoscopic sclerotherapy (EST) and band ligation (EBL). Endoscopic therapy is a local treatment that has no effect on the pathophysiological mechanisms that lead to portal hypertension and variceal rupture. However, a spontaneous decrease in HVPG occurs in around 30% of patients treated with either EST or EBL to prevent variceal rebleeding.
  Interventions: Device: Esophagogastroduodenoscope

INTERVENTIONS:
Device: Esophagogastroduodenoscope — Endoscopic therapies for varices aim to reduce variceal wall tension by obliteration of the varix. The two principal methods available for esophageal varices are endoscopic sclerotherapy (EST) and band ligation (EBL). Endoscopic therapy is a local treatment that has no effect on the pathophysiological mechanisms that lead to portal hypertension and variceal rupture. However, a spontaneous decrease in HVPG occurs in around 30% of patients treated with either EST or EBL to prevent variceal rebleeding.
  Other Names: EGD, upper GI endoscopy

SUMMARY:
Aim of this thesis is to predict the incidence of esophageal ulcer bleeding after endoscopic management of esophageal varices.

This study will be in the department of Tropical Medicine and Infectious Diseases, Tanta University, in at least six months in the period from august 2014 to march 2015 or until the target number of patients reached whichever is longer.

DETAILED DESCRIPTION:
Portal hypertension is a common clinical syndrome, defined by a pathologic increase in the portal venous pressure, in which the hepatic venous pressure gradient (HVPG) is increased above normal values (1-5 mmHg). In cirrhosis, portal hypertension results from the combination of increased intrahepatic vascular resistance and increased blood flow through the portal venous system.

Esophageal variceal bleeding is one of the most serious complications of portal hypertension, and represents a leading cause of death in patients with cirrhosis. Each bleeding episode is associated with a 30% mortality rate.

Endoscopic therapies for varices aim to reduce variceal wall tension by obliteration of the varix. The two principal methods available for esophageal varices are endoscopic sclerotherapy (EST) and band ligation (EBL). Endoscopic therapy is a local treatment that has no effect on the pathophysiological mechanisms that lead to portal hypertension and variceal rupture. However, a spontaneous decrease in HVPG occurs in around 30% of patients treated with either EST or EBL to prevent variceal rebleeding. EST consists of the injection of a sclerosing agent into the variceal lumen or adjacent to the varix, with flexible catheter with a needle tip, inducing thrombosis of the vessel and inflammation of the surrounding tissues. During active bleeding, sclerotherapy may achieve hemostasis, inducing variceal thrombosis and external compression by tissue edema. With repeated sessions, the inflammation of the vascular wall and surrounding tissues leads to fibrosis, resulting in variceal obliteration.

Furthermore, vascular thrombosis may induce ulcers that also heal, inducing fibrosis. There are technical variations in performing EST, such as type and concentration of the sclerosants, volume injected, interval between sessions, and number of sessions Endoscopic band ligation (EBL) is generally accepted as the treatment of choice for bleeding from esophageal varices. It has shown good results in terms of the control of the active bleeding, with few untoward effects.

Esophageal ulcerations ulcerations occur in the esophageal mucosa after all successful ligations. However, ulcers following Esophageal Variceal Ligation (EVL) are less severe than with ES.

Aim of this thesis is to predict the incidence of esophageal ulcer bleeding after endoscopic management of esophageal varices.

. This study will be in the department of Tropical Medicine and Infectious Diseases, Tanta University, in at least six months in the period from august 2014 to march 2015 or until the target number of patients reached whichever is longer.

The study include more than 224 patients who undergo endoscopic management of esophageal varices:

Methods:

All patients will be subjected to:

* full history taking.
* -complete clinical examination.
* -investigations for all groups: i) Complete Blood Count (CBC) ii) liver function tests iii) Kidney function tests. iv) ultrasound on abdomen and pelvis
* Upper endoscopy at day 0 , follow up endoscopy at day 14 and at 6months

End points:

1. ry end point:at 14 days to look for and characterize ulcer if any
2. ry end point: at 6months to look for general and local outcome of intervention

Inclusion criteria:

Patient with esophageal varices having upper GIT endoscopy

Exclusion criteria:

Patients having endoscopy with no esophageal varices (EVs)

ETHICAL CONSIDERATIONS Unexpected risks during the course of the research will be cleared to the participants and the ethical committee on time , thrombophlebitis may occur during taking blood sample, the investigators will use sterilized techniques during taking sample also bleeding from pinpoint needle track could happen , the investigators will do needle track ablation to avoid it. The investigators will use sterilized techniques during taking sample.

Informed consent will be taken and everyone will be given a coded number . Names will not be mentioned ,no pictures will be taken to any part of the body. Results of investigations will be collected, tabulated and statistically analyzed for scientific purposes only.

ELIGIBILITY:
Inclusion Criteria:

* Patient with esophageal varices having upper GIT endoscopy

Exclusion Criteria:

* Patients having endoscopy with no EVs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of esophageal ulcer bleeding after endoscopic management of esophageal varices. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Asem A Elfert, MD, Principal Investigator — Tanta Faculty of Medicine, Professor; Fat-heya E Assel, MD', Study Director — Tanta Faculty of Medicine, Professor; Ferial Elkalla, MD, Study Director — Tanta Faculty of Medicine, Professor; Galal Elkassas, MD, Study Director — Tanta Faculty of Medicine, Professor; Mohamed Elhendawy, Study Director — Dr.; Loai Mansour, Study Director — Dr.; Mohamed Rabei, Study Director — Dr.; Samah Mosaad, Study Director — Dr.; Ibrahim A Kabbash, MD, Study Director — Tanta Faculty of Medicine, Professor; Mohamed Elkassas, Study Director — Dr.; Islam S Ismail, Study Director — Dr.; Ibrahim Shebl, Study Director — Dr.
Locations (1):
- Tanta University Hospital, Tanta, Gharbia Governorate, Egypt

REFERENCES:
- [Result] Rigau J, Bosch J, Bordas JM, Navasa M, Mastai R, Kravetz D, Bruix J, Feu F, Rodes J. Endoscopic measurement of variceal pressure in cirrhosis: correlation with portal pressure and variceal hemorrhage. Gastroenterology. 1989 Mar;96(3):873-80. PMID 2783677
- [Result] Garcia-Tsao G, Groszmann RJ, Fisher RL, Conn HO, Atterbury CE, Glickman M. Portal pressure, presence of gastroesophageal varices and variceal bleeding. Hepatology. 1985 May-Jun;5(3):419-24. doi: 10.1002/hep.1840050313. PMID 3873388
- [Result] Cales P, Pascal JP. [Natural history of esophageal varices in cirrhosis (from origin to rupture)]. Gastroenterol Clin Biol. 1988 Mar;12(3):245-54. No abstract available. French. PMID 3286356
- [Result] de Franchis R. Endoscopy critics vs. endoscopy enthusiasts for primary prophylaxis of variceal bleeding. Hepatology. 2006 Jan;43(1):24-6. doi: 10.1002/hep.21026. No abstract available. PMID 16374843
- [Result] Garcia-Pagan JC, De Gottardi A, Bosch J. Review article: the modern management of portal hypertension--primary and secondary prophylaxis of variceal bleeding in cirrhotic patients. Aliment Pharmacol Ther. 2008 Jul;28(2):178-86. doi: 10.1111/j.1365-2036.2008.03729.x. Epub 2008 May 2. PMID 18462268
- [Result] Villanueva C, Lopez-Balaguer JM, Aracil C, Kolle L, Gonzalez B, Minana J, Soriano G, Guarner C, Balanzo J. Maintenance of hemodynamic response to treatment for portal hypertension and influence on complications of cirrhosis. J Hepatol. 2004 May;40(5):757-65. doi: 10.1016/j.jhep.2004.01.017. PMID 15094222
- [Result] Villanueva C, Colomo A, Aracil C, Guarner C. Current endoscopic therapy of variceal bleeding. Best Pract Res Clin Gastroenterol. 2008;22(2):261-78. doi: 10.1016/j.bpg.2007.11.012. PMID 18346683
- [Result] de Franchis R, Primignani M. Endoscopic treatments for portal hypertension. Semin Liver Dis. 1999;19(4):439-55. doi: 10.1055/s-2007-1007131. PMID 10643628
- [Result] Westaby D. Emergency and elective endoscopic therapy for variceal haemorrhage. Baillieres Clin Gastroenterol. 1992 Sep;6(3):465-80. doi: 10.1016/0950-3528(92)90033-b. No abstract available. PMID 1421595
- [Result] Villanueva C, Sancho-Poch F, Balanz Jea. Esophagic Histophathologic changes induced by variceal sclerosing therapy. Gastroenterol Hepatol 1990; 13: 15-19
- [Result] Helmy A, Hayes PC. Review article: current endoscopic therapeutic options in the management of variceal bleeding. Aliment Pharmacol Ther. 2001 May;15(5):575-94. doi: 10.1046/j.1365-2036.2001.00950.x. PMID 11328251
- [Result] Young MF, Sanowski RA, Rasche R. Comparison and characterization of ulcerations induced by endoscopic ligation of esophageal varices versus endoscopic sclerotherapy. Gastrointest Endosc. 1993 Mar-Apr;39(2):119-22. doi: 10.1016/s0016-5107(93)70049-8. PMID 8495829